CLINICAL TRIAL: NCT01358851
Title: A Prospective Comparator Controlled Randomized Exploratory Study on the Efficacy of LAS 41005 Compared to Cryotherapy in Subjects With Hyperkeratotic Actinic Keratosis
Brief Title: LAS41005 in Hyperkeratotic Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H 1005 6002 1007
Record Dates: First submitted 2011-05-02; First posted 2011-05-24 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Cryotherapy

ARMS (2):
- 1 (Experimental): Drug Las41005
  Interventions: Drug: LAS41005
- 2 (Other): Cryotherapy
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Cryotherapy — 1-2 times during the treatment time
  Arms: 2
Drug: LAS41005 — once daily
  Arms: 1

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of LAS 41005 compared to cryotherapy in subjects with moderate to severe hyperkeratotic actinic keratosis (punch biopsies).

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated written informed consent.
* Men and women aged between 18 and 85 years inclusive.
* Have a general good and stable health condition as confirmed by a physical examination and by medical history.
* Have at least 4 but not more than 10 clinically confirmed hyperkeratotic AK target lesions of moderate to severe intensity within the face/forehead or bald scalp
* Skin type I to IV according to Fitzpatrick's .
* Are free of any significant physical abnormalities (e.g., tattoos, dermatoses) in the potential treatment area that may cause difficulty with examination or final evaluation.
* Physical ability to apply the study preparation correctly and to follow the study restrictions and visit.
* Women of childbearing potential are allowed to participate in this study, only if they use a highly effective method of contraception

Main Exclusion Criteria:

* Have received treatment of AK within the treatment area (face / scalp) in the three months preceding this clinical trial.
* Have known hypersensitivity to the ingredients
* Are subjects under immunosuppressive therapy.
* Having coagulation defects which are inherited or acquired
* Have evidence of clinically significant, unstable medical conditions
* Have currently other malignant or benign tumors of the skin within the treatment area
* Subjects who have taken topical or systemic treatments that might interfere with the study end points, within a time window that is not allowed, or who are currently taking phenytoin, methotrexate or sulfonylurea.
* Subjects taking inhibitors of DPD (e.g. Brivudin, Sorivudin)
* Are known to be pregnant or lactating (currently or within the past 3 months).
* Have any dermatological disease in the treatment area or surrounding area that may be exacerbated by treatment
* Are currently or within the past 8 weeks participating in another clinical study.
* Have active chemical dependency or alcoholism as assessed by the investigator.
* Subject is institutionalized because of legal or regulatory order.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Histological status (AK diagnosis and grade) of one predefined target lesion | Screening and 8 weeks after last treatment
  Histological clearance at 8 weeks after end of treatment with LAS 41005, respectively 14 weeks after first cryotherapy. Histological Status will be measured by Histological Biopsy in order to confirm the diagnosis of AK and the grade.

SECONDARY OUTCOMES:
Total Actinic keratoses (AK)lesion count at each visit | day 1, day 21, day 42 and day 98.
  The clearance rate (complete/partial) of AK lesions (determined by clinical evaluation) in the treatment area (target areas A and B) will be measured by comparing the total AK lesion counts pre-treatment (on Day 1 before study treatment has been applied) with the lesion counts measured.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Rodríguez, Study Director — Almirall, S.A.
Locations (4):
- Germany (4):
  - Almirall investigative site 3, Dülmen
  - Almirall investigative site 1, Leipzig
  - Almirall investigative site 4, Soest
  - Almirall investigative site 2, Wuppertal

REFERENCES:
- [Derived] Simon JC, Dominicus R, Karl L, Rodriguez R, Willers C, Dirschka T. A prospective randomized exploratory study comparing the efficacy of once-daily topical 0.5% 5-fluorouracil in combination with 10.0% salicylic acid (5-FU/SA) vs. cryosurgery for the treatment of hyperkeratotic actinic keratosis. J Eur Acad Dermatol Venereol. 2015 May;29(5):881-9. doi: 10.1111/jdv.12702. Epub 2014 Sep 25. PMID 25257941